CLINICAL TRIAL: NCT01647724
Title: Experimentation of New Organizational Models of Cervical Cancer Screening Programs, Upon the Use of HPV Test as First Level: Evaluation of the Methodologies Proposed of the Use of Self-sampling Devices to Recover Non-responders.
Brief Title: New Methods of Distribution of a Self Sampler Kit for Cervical Cancer Screening
Acronym: NMDSS2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria Locale 4, Teramo (Other)
Responsible Party: Principal Investigator, Emma Altobelli, Responsable U.O. Epidemiology and Social Marketing, Azienda Sanitaria Locale 4, Teramo
Other Study IDs: NMD2TE
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-05

CONDITIONS: Cervical Cancer Cin Grade
Keywords: cervical cancer; prevention; screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — vaginal washings
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- control 1: standard recall letter to perform HPV test at the clinic
- Intervention 1: direct mailing of the self sampling device at home
- intervention 2: invitation to retire the self sampling device in local pharmacy

SUMMARY:
The opportunity of a home, self-collected sample, opens the chance to remove some of the barriers that may discourage women from participating to screening programmes or performing HPV (Human Papilloma Virus)-test. Self-sampling is less time consuming and invasive as compared with tests performed at a clinic. It allows for privacy, reduces discomfort and women know nobody would have to handle their body.

Study hypothesis: The use of a self-sampler may increase the recovery of non-responders women at cervical cancer screening.

DETAILED DESCRIPTION:
In a previous trial (ISRCTN96071600) the investigators tested on 2400 women, compliance with self sampler device (PantaRhei Devices, Zeist, the Netherlands).

With this study the investigators analyze the response to two channels of transmission of the device (a model of device easier, and less expensive than the previous), such as screening for colon cancer.

The shipment of the device at home and taking on a local pharmacy. Involving 15000 women non-responders to previous calls in five different screening programs in Italy (Rome, Bologna, Abruzzo region, Molise region, Veneto region).

ELIGIBILITY:
Inclusion Criteria:

All women (aged 35-64 years) non-responding to the screening invitation in the previous year and eligible for recall

Exclusion Criteria:

does not meet inclusion criteria

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Involving 15000 women non-responders to previous calls in five different screening programs in Italy (Rome, Bologna, Abruzzo region, Molise region, Veneto region).
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
performing a HPV test within 3 months since the recall letter | up to december 2012 (up to 3 months)

SECONDARY OUTCOMES:
How many of the women performing a test after intervention were never-screened or under-screened (last test more than 3 years before) | up to december 2012 (up to 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Altobelli, Prof., Study Director — AUSL4 Teramo - Italy
Locations (1):
- AUSL4 Teramo, Teramo, TE, Italy

REFERENCES:
- [Derived] Giorgi Rossi P, Fortunato C, Barbarino P, Boveri S, Caroli S, Del Mistro A, Ferro A, Giammaria C, Manfredi M, Moretto T, Pasquini A, Sideri M, Tufi MC, Cogo C, Altobelli E; HPV Self-sampling Italian Working Group. Self-sampling to increase participation in cervical cancer screening: an RCT comparing home mailing, distribution in pharmacies, and recall letter. Br J Cancer. 2015 Feb 17;112(4):667-75. doi: 10.1038/bjc.2015.11. Epub 2015 Jan 29. PMID 25633037